CLINICAL TRIAL: NCT01474226
Title: Application of the Indicator Amino Acid Oxidation Technique for the Determination of Metabolic Availability of Lysine From Cooked Rice Protein in Adult Men
Brief Title: Metabolic Availability of Lysine From Rice
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Dr. Paul Pencharz, Professor of Paediatrics and Nutritional Sciences (Emeritus) University of Toronto, Senior Scientist Research Institute,The Hospital for Sick Children, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0019850580; CIHR, grant MT10321 (Other Grant/Funding Number: CIHR, grant MT10321)
Record Dates: First submitted 2011-11-10; First posted 2011-11-18 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Adults
Keywords: lysine; rice; bioavailability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lysine Amino Acid (Experimental)
  Interventions: Dietary Supplement: Amino Acid Crystalline Lysine Amino Acid Mix; Dietary Supplement: Cooked Rice containing Lysine

INTERVENTIONS:
Dietary Supplement: Amino Acid Crystalline Lysine Amino Acid Mix — crystalline lysine from AA MIX (20, 40, and 60% of the mean lysine requirement of 35 mg/kg/d) Lysine will be given in the form of L-Lysine-HCl, Sigma-Aldrich Brand.
Dietary Supplement: Cooked Rice containing Lysine — Lysine (20,40 and 60 % of the mean lysine requirement) from Cooked Rice

SUMMARY:
The purpose of this study is to investigate the digestibility of the amino acid lysine in cooked rice in adult men using stable isotope technique.

DETAILED DESCRIPTION:
The investigators objective is to determine the metabolic availability (MA) of lysine in cooked white rice protein using the indicator amino acid oxidation (IAAO) technique. Five men will receive graded levels (20, 40, and 60, and 70%) of the lysine requirement of 35 mg/kg/d as a crystalline AA mixture,and cooked rice protein (20, 40 and 60%), respectively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adult males (18 to 50years old)

Exclusion Criteria:

* A history of recent weight loss or illness
* Use of any medication at the time of entry into the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Metabolic Availability of lysine | Baseline
  3 breath samples will be taken to provide a baseline F13CO2 measurement (Level of phenylalanine oxidation). Breath samples will be collected and analyzed for 13CO2 enrichment.
Metabolic Availability of lysine | 15 min after intake of the fourth hourly meal (before tracer infusion))
  3 breath samples will be taken to provide a baseline F13CO2 measurement (Level of phenylalanine oxidation). Breath samples will be collected and analyzed for 13CO2 enrichment.
Metabolic Availability of lysine | 30 min after intake of the fourth hourly meal (before tracer infusion))
  3 breath samples will be taken to provide a baseline F13CO2 measurement (Level of phenylalanine oxidation). Breath samples will be collected and analyzed for 13CO2 enrichment.
Metabolic Availability of lysine | 45 min after intake of the fourth hourly meal (before tracer infusion))
  3 breath samples will be taken to provide a baseline F13CO2 measurement (Level of phenylalanine oxidation). Breath samples will be collected and analyzed for 13CO2 enrichment.

SECONDARY OUTCOMES:
Metabolic Availability of Lysine | Post Tracer Infusion (between 150 and 240 min of tracer infusion)
  4 breath samples will be taken to provide F13CO2 measurement (Level of phenylalanine oxidation).Breath samples will be collected and analyzed for 13CO2 enrichment.

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Pencharz, MD, PhD, Principal Investigator — The Hospital for Sick Children, Toronto, Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Prolla IR, Rafii M, Courtney-Martin G, Elango R, da Silva LP, Ball RO, Pencharz PB. Lysine from cooked white rice consumed by healthy young men is highly metabolically available when assessed using the indicator amino acid oxidation technique. J Nutr. 2013 Mar;143(3):302-6. doi: 10.3945/jn.112.166728. Epub 2013 Jan 16. PMID 23325920